CLINICAL TRIAL: NCT02973191
Title: A Phase 2, Open-label, Multiple Cohort, Single-arm, Multi-center Trial to Determine the Safety, Feasibility and Efficacy of JCAR015 in Adult Subjects With B-cell Acute Lymphoblastic Leukemia.
Brief Title: A Study to Determine Safety, Feasibility and Efficacy of JCAR015 in Adult Subjects With B-Cell Acute Lymphoblastic Leukemia
Acronym: ORBIT
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Development of JCAR015 has been discontinued. No subjects were enrolled/treated under protocol JCAR015-ALL-001
Sponsor: Celgene (Industry)
Collaborators: Juno (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: JCAR015-ALL-001
Record Dates: First submitted 2016-11-22; First posted 2016-11-25 (Estimated); Last update posted 2017-04-10 (Actual); Status verified 2017-04

CONDITIONS: Precursor Cell Lymphoblastic Leukemia-Lymphoma
Keywords: Leukemia; B-Cell Acute Lymphoblastic Leukemia; JCAR015
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia; Burkitt Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- JCAR015 administration (Experimental): Single dose of 1.0-3.0 mg/m^2 IV cyclophosphamide, JCAR015 Dose 1 1x10^6 Tcells/kg, JCAR015 Dose 2 3x10^6 Tcells/kg
  Interventions: Drug: JCAR015

INTERVENTIONS:
Drug: JCAR015

SUMMARY:
This is a single-arm, multi-center, open-label, Phase 2 study to determine the efficacy and safety of JCAR015 in adult subjects with B-cell ALL. The study is divided into two sequential parts, Part A and Part B; subjects will be screened and will provide informed consent before initiating any study procedures in Part A of the study.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18 years at the time of signing the informed consent form
2. Subject must understand and voluntarily sign an Informed consent form (ICF) prior to any study-related assessments/procedures being conducted
3. Subject is willing and able to adhere to the study visit schedule and other protocol requirements
4. Diagnosis of B-cell Acute Lymphoblastic Leukemia (ALL)
5. Evidence of CD19 expression via flow cytometry (peripheral blood or bone marrow) or immunohistochemistry (bone marrow biopsy)
6. Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2
7. No contraindications to cyclophosphamide. This includes subjects with:

   * hypersensitivity to cyclophosphamide, any of its metabolites
   * acute infections
   * bone marrow aplasia or bone marrow depression prior to treatment
   * urinary tract infection
   * acute urothelial toxicity from cytotoxic chemotherapy or radiation therapy
   * urinary outflow obstruction
   * obstruction
8. Adequate organ function, defined as:

   a. Serum creatinine ≤ 1.5 × age-adjusted upper limit of normal (ULN) OR calculated creatinine clearance (Cockcroft and Gault) > 30 mL/min/1.73 m2 b. Alanine aminotransferase (ALT) ≤ 5 × ULN and direct bilirubin < 2.0 mg/dL (or < 3.0 mg/dL for subjects with leukemic infiltration of the liver) c. Adequate pulmonary function, defined as ≤ Grade 1 dyspnea and oxygen saturation (SaO2) ≥ 92% on room air d. Adequate cardiac function, defined as left ventricular ejection fraction (LVEF) ≥ 40% as assessed by echocardiogram (ECHO) or multiple uptake gated acquisition (MUGA) performed within 1 month of signing the informed consent form
9. Adequate central or peripheral vascular access for leukapheresis procedure. For subjects requiring central venous catheter (CVC) placement, a surgical consultation indicating subject eligibility for CVC placement is sufficient for enrollment.
10. Subjects must agree to not donate blood, organs, sperm or semen, and egg cells for usage in other individuals without recipient knowledge about exposure to a genetically modified organ by the donor and having been informed about the potential risks associated with it at any point after receiving JCAR015 infusion.
11. Females of childbearing potential (FCBP1) must:

    a. Have two negative pregnancy tests as verified by the Investigator (one negative serum beta human chorionic gonadotropin (ß-hCG) pregnancy test result within 7 days prior to the first dose of cytoreductive chemotherapy (Part A screening evaluation), and one negative serum or urine pregnancy test at the Part B screening evaluation prior to first JCAR015 infusion). She must agree to have another pregnancy test 90 days post final JCAR015 dose. This applies even if the subject practices true abstinence2 from heterosexual contact.

    b. Either commit to true abstinence2 from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use, and be able to comply with, effective contraception without interruption. Contraception methods must include 1 highly effective and 1 additional effective (barrier) method of contraception from at least 28 days prior to JCAR015 initial infusion and during the study therapy including dose interruptions. Cessation of contraception after this point should be discussed with a responsible physician. Note: Highly effective methods are defined as those that result in a low failure rate (ie, less than 1% per year) when used consistently and correctly. The following are examples of highly effective and additional effective methods of contraception:

    - Intrauterine device (IUD)

    - Hormonal (birth control pill, injections, implants)

    - Tubal ligation

    - Partner's vasectomy

    - Male Condom (additional effective method)

    - Diaphragm (additional effective method)

    - Cervical Cap (additional effective method) c. Agree to abstain from breastfeeding during study participation and for at least 90 days after the last dose of JCAR015.

    d. Agree to use highly effective methods of contraception during the entire study period (Part A through 12 months after the final JCAR015 infusion).
12. Males who have partners of childbearing potential must agree to use an effective barrier contraceptive method during the entire study period (Part A through 12 months after the final JCAR015 infusion).

Additional Cohort Specific Inclusion Criteria

Inclusion Criteria (Cohorts 1-4) 1. Relapsed or refractory disease, defined as:

1. First bone marrow relapse (prior Complete response (CR) duration < 18 months) or any subsequent bone marrow relapse from Complete response (CR), OR
2. Any bone marrow relapse after allogeneic hematopoietic stem cell transplant (HSCT); subjects must be at least 2 months from HSCT at the time of signing the informed consent form and off immunosuppressant medication for at least 1 month at the time of signing the informed consent form (with the exception of low-dose steroids (≤ 20 mg prednisone or equivalent), and have no Graft versus host disease (GVHD), OR
3. Refractory Acute Lymphoblastic Leukemia (ALL), defined by not having achieved a Complete response (CR) or Complete response with incomplete peripheral blood count recovery (CRi) after two attempts at remission induction using standard chemotherapy regimens, OR
4. Philadelphia chromosome positive (Ph+) B-cell ALL if subjects are intolerant to, or ineligible for, Tyrosine kinase inhibitor (TKI) therapy, or have progressed after at least one line of TKI therapy.

   2. Bone marrow with morphological evidence of disease (≥ 5% blasts by morphology).

   Inclusion Criteria [Ph(+) (Cohort 3)] All subjects must meet Inclusion criteria described for Cohort 1.

   Inclusion Criteria (Cohort 4 only) 1. Eligible for Cohorts 1-3 but investigator has decided to administer blinatumomab as standard ALL therapy rather than other alternatives listed after leukapheresis but prior to part B of therapy Inclusion Criteria (MRD Positive+ [Cohort 5])

   Inclusion criteria as for Cohorts 1 and 2, with the exception of:

   1. Bone marrow without morphological evidence of disease characterized as ≤ 5% blasts by morphology, but with MRD detected by flow cytometry, or qPCR at a frequency of ≥ 1 x 10-4 following standard of care induction and consolidation therapy in CR1 or in any subsequent CR
   * For subjects in whom MRD has been followed only by flow cytometry, a nucleic acid sample of the leukemia blasts of sufficient quality must be available to generate realtime quantitative PCR (RQ-PCR) primers.

   4.2.2. Inclusion Criteria (Part B)

   1. Completion of Part A and successful generation of a JCAR015 cell product 2. Results from bone marrow examination following Part A:

<!-- -->

1. Group 1: Morphological evidence of disease (≥ 5% blasts by morphology)
2. Group 2: Morphologic complete remission (bone marrow with < 5% blasts) with or without blood count recovery (CR or CRi) or a hypoplastic, aplastic, or "recovery" marrow at Day 42 of Part A 3. Eastern Cooperative Oncology Group (ECOG) performance status between 0 and 2 4. Adequate organ function, defined as:

<!-- -->

1. Serum creatinine ≤ 1.5 × age-adjusted ULN OR calculated creatinine clearance
2. (Cockcroft and Gault) > 30 mL/min/1.73 m2
3. ALT ≤ 5 × ULN (or ≤ 8 × ULN for subjects with leukemic infiltration of the liver) and direct bilirubin < 2.0 mg/dL (or < 3.0 mg/dL for subjects with leukemic infiltration of the liver)
4. Adequate pulmonary function, defined as ≤ Grade 1 dyspnea and SaO2 ≥ 92% on room air 5. Females of childbearing potential and males who have partners of childbearing potential follow the same inclusion criteria as Part A.

Exclusion Criteria:

1. Isolated extramedullary disease relapse
2. Concomitant genetic syndrome such as Fanconi anemia, Kostmann syndrome, Shwachman syndrome, or any other known bone marrow failure syndrome
3. Burkitt's lymphoma/leukemia or chronic myelogenous leukemia (CML) lymphoid blast crisis (p210 BCR-ABL+)
4. Prior malignancy, unless treated with curative intent and with no evidence of active disease present for > 5 years before signing the informed consent form, with the following exceptions:

   a. Subjects with Stage I breast cancer that has been completely and successfully treated, requiring no therapy or only anti-hormonal therapy b. Subjects with T1N0M0 or T2N0M0 colorectal cancer who have been completely and successfully resected and who are disease-free for > 2 years prior to screening c. Subjects with indolent prostate cancer, defined as clinical stage T1 or T2a, Gleason score ≤ 6, and prostate-specific antigen (PSA) < 10 ng/mL, requiring no therapy or only anti- hormonal therapy d. Subjects with a history of basal cell or squamous cell carcinoma of the skin, or carcinoma in situ of the cervix, fully resected, and with no evidence of active disease
5. Treatment with any prior gene therapy product
6. Active hepatitis B, active hepatitis C, or any human immunodeficiency virus (HIV) infection at the time of signing the informed consent form
7. Systemic fungal, bacterial, viral, or other infection that is not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment) at the time of signing the informed consent form
8. Presence of Grade II-IV (Glucksberg) or B-D (IBMTR) acute or extensive chronic GVHD at the time of signing the informed consent form
9. Active C S involvement by malignancy, defined as CNS-3 per NCCN guidelines. Subjects with a history of Central nervous system (CNS) disease that has been effectively treated (defined as one documented negative CSF evaluation within 1 month prior to signing the informed consent form) will be eligible
10. History of any one of the following cardiovascular conditions within the past 6 months of signing the informed consent form: Class III or IV heart failure as defined by the New York Heart Association (NYHA), cardiac angioplasty or stenting, myocardial infarction, unstable angina, or other clinically significant cardiac disease
11. History or presence of clinically relevant CNS pathology such as epilepsy, generalized seizure disorder, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis
12. Participation in an investigational research study using an investigational agent within 30 days of signing the informed consent form, with the exception of investigational antiinfective agents (eg, antibacterial, antifungal, antiviral)
13. History of treatment with a murine-derived biological product (unless subject has been shown to be negative for human anti-mouse antibodies [HAMA] prior to or during screening). Prior use of blinatumomab is permitted (provided there is evidence of CD19 expression per Part A Inclusion Criterion #4). Chimeric biological products (eg, rituximab) are not considered murine for the purpose of this protocol.
14. Pregnant or nursing (lactating) women
15. Use of prohibited medications:

    a. Steroids: Therapeutic doses of corticosteroids (defined as > 20 mg/day prednisone or equivalent) are prohibited within 7 days prior to leukapheresis. Physiologic replacement dosing of steroids (≤ 12 mg/m2/day hydrocortisone or equivalent [≤ 3 mg/m2/day prednisone or ≤ 0.45 mg/m2/day dexamethasone]) is allowed. Topical steroids and intrathecal steroids for CNS relapse prophylaxis are permitted.

    b. Allogeneic cellular therapy: Donor lymphocyte infusions (DLI) are prohibited within 4 weeks prior to leukapheresis c. GVHD therapies: Any drug used for GVHD within 4 weeks prior to leukapheresis, eg, calcineurin inhibitors, methotrexate or other chemotherapeutics, mycophenolate mofetil, rapamycin, thalidomide, immunosuppressive antibodies (such as anti-CD20 [rituximab], anti-TNFα, anti-IL-6, or anti-IL-6R) d. Chemotherapies: Salvage chemotherapy (eg, cytosine arabinoside > 100 mg/m2/day, anthracyclines, and cyclophosphamide) must be stopped at least 1 week prior to leukapheresis
16. Treatment with alemtuzumab within 6 months prior to leukapheresis, or treatment with clofarabine or cladribine within 3 months prior to leukapheresis
17. Uncontrolled medical, psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol, as judged by the Investigator; or subject unwillingness or inability to follow the procedures required in the protocol 4.3.2. Exclusion Criteria (Part B)

Subjects must not meet any of the following criteria prior to Part B to be considered eligible:

1. Systemic fungal, bacterial, viral, or other infection that is not controlled (defined as exhibiting ongoing signs/symptoms related to the infection and without improvement, despite appropriate antibiotics or other treatment)
2. Active CNS involvement by malignancy, defined as CNS-3 per NCCN guidelines. Subjects with a history of CNS disease that has been effectively treated (defined as one documented negative CSF evaluation within 1 month prior to signing the informed consent form) will be eligible
3. Presence of clinically relevant CNS pathology such as epilepsy, generalized seizure disorder, paresis, aphasia, stroke, severe brain injuries, dementia, Parkinson's disease, cerebellar disease, organic brain syndrome, or psychosis
4. Presence of Grade II-IV (Glucksberg) or B-D (IBMTR) acute or extensive chronic GVHD
5. Use of prohibited medications
6. Female subjects that have a positive serum or urine pregnancy test, or are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-12-20 (Estimated); Primary Completion 2019-06-25 (Estimated); Study Completion 2021-01-24 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to 6 months
  The primary efficacy endpoint (for Cohorts 1-4) is ORR as determined by an Independent Review Committee (IRC). The ORR is, defined as proportion of subjects with a best overall response of Complete response (CR) or Complete response with incomplete peripheral blood count recovery (CRi) from 28 days through 6 months after the final infusion of JCAR015 or the start of receiving another anti-cancer therapy whichever comes first.
Minimal residual disease (MRD) | Up to 90 days
  Evaluate the proportion of subjects who achieve a MRD negative complete response (CR) and the duration of MRD negative status, if achieved, after JCAR015 administration.

SECONDARY OUTCOMES:
Adverse Events (AEs) | Up to 2 years
  Number participants with adverse events
Duration of Minimal residual disease (MRD) response | Up to 24 months
  Time from Minimal Residual Disease (MRD) response until MRD recurrence, morphologic relapse, or death
Relapse-free survival (RFS) | Up to 24 months
  Relapse-free survival (RFS) is defined as the interval from the first documentation of complete response (CR) or Complete response with incomplete peripheral blood count recovery (CRi) to the earlier date of relapse or death due to any cause.
Event-free survival (EFS) | Up to 24 months
  Is defined as the time from the date of the first JCAR015 infusion to death from any cause, relapse, or treatment failure, whichever occurs first
Overall survival (OS) | Up to 24 months
  Is defined as the time from the date of the first JCAR015 infusion to date of death due to any reason
Percent Minimal residual disease (MRD) negative | Up to 24 months
  Percentage of subjects who achieve CR or CRi with an MRD-negative bone marrow, as assessed by IgH gene sequencing (or BCR-ABL qPCR or flow cytometry for Ph(+) ALL subjects)
Depth of Minimal residual disease (MRD) response | Up to 24 months
  Improvement of response in patients with MRD+ ALLL
Duration of remission (DOR) | Up to 24 months
  Is defined as the interval from the first documentation of CR or CRi to the earlier date of relapse or death due to ALL. The first documentation of CR or CRi is defined as the latest of all dates of required measurements to establish the response. Duration of remission (DOR) will be evaluated based on the IRC evaluations for subjects who achieve a CR or CRi.
Pharmacokinetics - Cmax | Up to 24 months
  Maximum observed concentration in plasma
Pharmacokinetics- Tmax | Up to 24 months
  Time to reach maximum observed concentration in plasma
Pharmacokinetics - AUC | Up to 24 months
  Area under the plasma concentration-time curve

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hasskarl, MD, Study Director — Celgene Corporation
Locations (18):
- Universitair Ziekenhuis Gent, Ghent, Belgium
- France (2):
  - University de Lille, Lille
  - Hopital Saint Louis, Paris
- Germany (6):
  - University of Cologne, Cologne
  - Universitaetsklinikum Carl Gustav Carus an der Technischen Universitaet Dresden, Dresden
  - Universitatsklinikum Frankfurt, Frankfurt
  - University of Munich Grosshadern, Grosshadern Campus
  - University of Leipzig, Leipzig
  - Universitaetsklinikum Ulm, Ulm
- Italy (4):
  - USC Ematologia, Azienda Ospedaliera Papa Giovanni XXIII, Bergamo
  - Istituto Clinico Humanitas - Istituti di Ricovero E Cura A Carattere Scientifico (IRCSS), Milan
  - Universita La Sapienza, Roma
  - Azienda Ospedaliera Citta della Salute e della Scienza di Torino, Torino
- Spain (2):
  - ICO-Hospital Germans Trias i Pujol, Barcelona
  - Hospital Universitario de Salamanca, Salamanca
- Chuv Bh-04, Lausanne, Switzerland
- United Kingdom (2):
  - Bristol Royal Infirmary, University of Bristol Foundation Trust, Bristol
  - UCL Cancer Institute, London